CLINICAL TRIAL: NCT02514967
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 3 Study to Evaluate the Efficacy and Safety of Blisibimod Administration in Subjects With Systemic Lupus Erythematosus With or Without Nephritis
Brief Title: CHABLIS7.5: A Study of the Efficacy and Safety of Subcutaneous Blisibimod in Subjects With Systemic Lupus Erythematosus With or Without Nephritis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study halted prematurely and will not resume. Subjects were seen until February 2017
Sponsor: Anthera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AN-SLE3343
Record Dates: First submitted 2015-07-31; First posted 2015-08-04 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE; Lupus; Lupus Erythematosus, Systemic; Autoimmune Diseases; A-623; Blisibimod; Nephritis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases; Nephritis | interventions — AMG623 peptibody

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Blisibimod (Experimental)
  Interventions: Drug: Blisibimod
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Blisibimod — Administered via subcutaneous injection once per week
  Arms: Blisibimod
Drug: Placebo — Administered via subcutaneous injection once per week
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy of blisibimod as measured by a composite responder index in subjects who, despite corticosteroid use, continue to have seropositive, clinically-active Systemic Lupus Erythematosus (SLE) as defined by SELENA-SLEDAI score ≥10, and positive for anti-double stranded DNA and low complement (C3 or C4).

ELIGIBILITY:
Inclusion Criteria:

* Fulfill at least 4 diagnostic criteria for SLE defined by American College of Rheumatology
* Active SLE disease as defined by SELENA-SLEDAI score ≥10 despite on-going stable corticosteroid therapy
* Positive for anti-double stranded DNA (anti-dsDNA) and low complement
* Subjects with stable nephritis may be enrolled
* 18 years of age or older

Exclusion Criteria:

* Severe active central nervous system lupus
* Malignancy within past 5 years
* Known to be positive for HIV and/or positive at the screening visit for hepatitis B, or hepatitis C
* Comorbidities that would interfere with evaluations of study drug effect
* Active infection requiring hospitalization or treatment with parenteral antibiotics within the past 60 days or history of repeated herpetic viral infections
* History of active tuberculosis or a history of tuberculosis infection
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Proportion of responders to the SRI-6 composite responder index | 52 Weeks

SECONDARY OUTCOMES:
Time to first severe SLE flare | Baseline through 52 weeks
Change in the number of actively tender or swollen joints and in mucocutaneous disease activity | 52 Weeks
Change in proteinuria from baseline | Week 52
Proportion of subjects able to reduce oral steroid dose to ≤ 7.5 mg | Baseline through 52 weeks
Proportion of subjects with improved patient-reported outcomes | Week 52
Time to treatment failure | Through week 52
Change from baseline in B cell counts, anti-dsDNA, C3, C4 | Through week 52
Number of adverse events | Through week 52

OTHER OUTCOMES:
Occurrence of renal flare in subjects with renal manifestations at baseline | 52 Weeks

CONTACTS AND LOCATIONS:
Locations (3):
- Georgia (3):
  - Investigator Site 004, Tbilisi
  - Investigator Site 001, Tbilisi
  - Investigator Site 002, Tbilisi

REFERENCES:
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069